CLINICAL TRIAL: NCT06182085
Title: Randomised, Double-blind, Placebo-controlled Study to Assess Safety and Efficacy of PRI-002 in Patients With MCI to Mild Dementia Due to Alzheimer's Disease (AD) (PRImus-AD)
Brief Title: Study to Assess Safety and Efficacy of PRI-002 in Patients With MCI to Mild Dementia Due to Alzheimer's Disease (AD)
Acronym: PRImus-AD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PRInnovation GmbH (Industry)
Collaborators: Priavoid (Unknown); Federal Agency for Disruptive Innovation - SPRIN-D (Unknown); Julius Clinical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRI-002-004
Record Dates: First submitted 2023-11-29; First posted 2023-12-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment Due to Alzheimer's Disease; Alzheimer's Disease, Early Onset
Keywords: PRI-002; PRImus-AD; Clinical Dementia Rating Sum of Boxes (CDR-SB); Prodromal Alzheimer's disease; Mild Alzheimer's disease dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Daily oral administration of 3 capsules in the morning and evening.
  Interventions: Drug: Placebo
- PRI-002, dosage arm 1 (Experimental): Daily oral administration of 3 capsules in the morning and evening, lower dose.
  Interventions: Drug: PRI-002
- PRI-002, dosage arm 2 (Experimental): Daily oral administration of 3 capsules in the morning and evening, higher dose.
  Interventions: Drug: PRI-002

INTERVENTIONS:
Drug: PRI-002 — Oral administration
  Other Names: Contraloid
  Arms: PRI-002, dosage arm 1; PRI-002, dosage arm 2
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is the most common form of dementia. In the brains of people with AD, certain small substances stick together. This leads to changes in thinking and behaviour. The company PRInnovation is developing a new treatment for Alzheimer's disease, called PRI-002. It is thought that PRI-002 can cut the sticked substances back into small pieces. That would reduce the effects of Alzheimer's disease. In the current study the investigators examine whether PRI-002 is safe and effective in participants with mild cognitive impairment (MCI) or mild dementia due to AD.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive neurodegenerative disorder and the most common form of dementia. The post-mortem pathology of AD is mainly characterised by neurodegeneration as well as extracellular amyloid plaques and intracellular neurofibrillary tangles. Research suggests that the amyloid-β-peptide (Aβ) aggregation plays a major role in the development of AD, while Aβ oligomers are thought to be the most toxic species. Therefore, various strategies to develop AD therapeutics address Aβ and some examples include trying to reduce its formation, inhibit its aggregation to fibrils or enhancing its clearance.

PRI-002 is being investigated as a possible treatment for cognitive impairment due to AD. PRI-002 is an all D-amino acid peptide (all-D-peptide) consisting of a rationally designed primary structure, resulting in efficient removal of Aβ oligomers. PRI-002 specifically aims to eliminate neurotoxic Aβ oligomers by disassembling prion-like behaving Aβ oligomers into non-toxic Aβ monomer units. This therapeutic principle is new and unique and differs from that of other amyloid related drug candidates currently in clinical development, which aim to increase the degradation rate of different Aβ species.

The current trial is a Phase 2 proof-of-concept study to further investigate the safety and efficacy of PRI-002 in patients with mild cognitive impairment (MCI) or mild dementia due to AD.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent obtained from the subject and study companion in accordance with applicable regulations.
2. Male or female, aged 55 to 80 years, inclusive.
3. For female subjects: not being of child-bearing potential. This is defined as either permanently sterilised (via hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or postmenopausal (defined as no menses for 12 months without an alternative medical cause).

   For male subjects who are sexually active with women of child-bearing potential: agreeing to use acceptable contraception (using a condom or having demonstrated successful vasectomy) and not donate sperm from Screening until 12 weeks after the last dose of study treatment.
4. Body mass index (BMI) between 18.5 and 30.0 kg/m2, inclusive.
5. Diagnosed with MCI due to AD or mild dementia due to AD, according to the NIA-AA criteria.
6. MMSE score of 22 to 30, inclusive.
7. Repeatable battery for the assessment of neuropsychological status - delayed memory index (RBANS-DMI) score ≤85.
8. CDR global score of 0.5 or 1 with a memory score ≥0.5.
9. Confirmation of AD diagnosis, by

   * CSF biomarker profile reflecting AD, according to NIA-AA, or
   * existing positive amyloid positron emission tomography (PET) evidence.
10. Fluency in local language and evidence of adequate intellectual functioning in the opinion of the investigator.
11. Having a reliable informant or caregiver who is willing and able to act as the study companion throughout the duration of the subject's participation. The subject and the study companion must have frequent interaction (defined as a minimum of 6 hours/week on average) according to subject's report.

Exclusion Criteria:

1. Unable to give informed consent in accordance with applicable regulations.
2. Diagnosed with moderate or severe dementia due to AD according to NIA-AA.
3. History or evidence of any other central nervous system (CNS) disorder(s) that could be interpreted as a cause of cognitive impairment or dementia.
4. History of known or suspected seizures, loss of consciousness, or significant head trauma within 2 years before Screening.
5. History of known or suspected stroke or transient ischaemic attack (TIA) within 2 years before Screening.
6. Evidence of other clinically significant lesions on brain MRI (Fazekas score 3).
7. History or presence of clinically evident cerebrovascular disease (diagnosis of possible, probable, or definite vascular dementia).
8. Other significant pathological findings on brain MRI (for example more than 10 microhaemorrhages or a single macrohaemorrhage >10 mm at the greatest diameter).
9. Unstable medical, neurological, or psychiatric condition, or presence of major depressive episode at Screening.
10. Life-time history of schizophrenia or history of uncontrolled bipolar disorder within 5 years before Screening.
11. Having a bleeding disorder that is not under adequate control (defined as a platelet count <50000 or international normalised ratio [INR] >1.5). Participants who are on anticoagulant therapy (for example, warfarin), should have their anticoagulant status optimised and be on a stable dose for 30 days before Screening. Anticoagulant therapy (e.g., clopidogrel bisulfate, carbasalate calcium 100 mg/day, or aspirin 325 mg/day or less) is permitted provided this therapy does not represent a contraindication for a lumbar puncture and CSF sampling (if CSF sampling is required in the absence of historical PET evidence).
12. Having significant kidney disease as indicated by either of the following:

    * Creatinine clearance (eGFR) ≤30 mL/min/1.73m2) as estimated using the modification of diet in renal disease (MDRD) method, or
    * Creatinine ≥2 mg/dL.
13. Having impaired hepatic function as indicated by aspartate amino transferase (AST) or alanine amino transferase (ALT) >3-fold the upper limit of normal (ULN), or total bilirubin >2-fold ULN, at Screening.
14. Known to be human immunodeficiency virus (HIV) positive.
15. Known to be hepatitis C or chronic hepatitis B positive.
16. Having any other clinically significant abnormalities in physical examination, vital signs, laboratory tests, MRI, or ECG at Screening or Baseline which in the opinion of the investigator requires further investigation or treatment or which may interfere with study procedures or safety.
17. Use of licensed symptomatic AD medication for less than 90 days or at a non-stable dose over the past 90 days at Baseline (for example acetylcholinesterase inhibitors, memantine, ginkgo).
18. Use of anti-Aβ monoclonal antibody therapy at Baseline.
19. Treatment with one of the following substances:

    1. Typical antipsychotic or neuroleptic medication within 90 days before Screening (except for

       ≤1 mg risperidon, and ≤300 mg quetiapin).
    2. Chronic use of opiates or opioids (including long-acting opioid medication) within 90 days before Screening.
    3. Stimulant medications (amphetamine, methylphenidate preparations, or modafinil) within 30 days before Screening.
    4. Chronic use of benzodiazepines, barbiturates, or hypnotics within 90 days before Screening.
20. Contraindication to MRI. Patients with MRI compatible pacemakers may be allowed to enter the study.
21. Prior or current participation in a clinical trial testing active immunisation against Aβ or tau.
22. Participation in a clinical trial and having taken at least 1 dose of the investigational medicinal product (IMP), within 5 times the IMP half-life time before Baseline, unless confirmed as having been on placebo.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple doses of PRI-002 in subjects with MCI or mild dementia due to AD, based on incidence of drug-related adverse events (AEs). | Baseline to week 48.
  Percentage of subjects with at least 1 drug- related AE or drug-related serious adverse event (SAE) between Baseline and Week 48.
To evaluate the efficacy of multiple doses of PRI-002 in subjects with MCI or mild dementia due to AD, based on the Clinical Dementia Rating - Sum of Boxes (CDR-SB). | Baseline to week 48.
  Change from Baseline to Week 48 in global outcome as measured by CDR-SB.

SECONDARY OUTCOMES:
To evaluate safety and tolerability of multiple doses of PRI-002 in subjects with MCI or mild dementia due to AD, based on AEs, amyloid related imaging abnormalities oedema (ARIA-E) and haemosiderin (ARIA-H), and treatment discontinuations due to AEs. | Through study completion up to 96 weeks.
  Percentage of subjects with AEs and SAEs from Baseline until End of Study (EoS).
To evaluate clinical outcome measures of multiple doses of PRI-002 in subjects with MCI or mild dementia due to AD. | Through study completion up to 48 weeks.
  Change from Baseline to Week 48 of:
  Alzheimer's disease cooperative study - activities of daily living inventory (ADCS-ADL), Alzheimer disease assessment scale - cognitive subscale, 13 tests (ADAS-Cog 13)
To evaluate clinical outcome measures of multiple doses of PRI-002 in subjects with MCI or mild dementia due to AD. | Baseline to study completion.
  Change from Baseline to study completion of: CDR-SB, ADCS-ADL, ADAS-Cog 13
To evaluate clinical outcome measures and biomarkers of multiple doses of PRI-002 in subjects with MCI or mild dementia due to AD. | Baseline to study completion.
  Change from Baseline to EoT of: Mini mental state examination (MMSE) scores, Cerebrospinal fluid (CSF) concentrations of AD-related biomarkers including, but not limited to, ratio Aβ 1-42/1-40, p-tau, t-tau, Aβ oligomers, and tau oligomers, Plasma concentrations of AD-related biomarkers including, but not limited to, ratio Aβ 1-42/1-40, p-tau, t-tau, neurofilament light chain (NfL), glial fibrillary acidic protein (GFAP), and Aβ oligomers, Correlations between changes in CSF and plasma biomarkers and clinical changes (CDR-SB, ADCS-ADL, ADAS-Cog 13, MMSE)
To follow drug levels of PRI-002 during multiple doses of PRI-002 in subjects with MCI or mild dementia due to AD. | Through study completion up to 96 weeks.
  PRI-002 plasma concentrations over time.
To evaluate the correlation between PRI-002 exposure and efficacy and the correlation between PRI-002 exposure and safety in subjects with MCI or mild dementia due to AD. | Through study completion up to 96 weeks.
  Correlations between PRI-002 plasma concentrations and clinical changes (CDR-SB, ADCS-ADL, ADAS-Cog 13, MMSE) and safety endpoints (AEs and SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Tischler, Dr., Study Chair — PRInnovation
Locations (38):
- Czechia (7):
  - Neuro Health Centrum ltd., Brno
  - NeuropsychiatrieHK, s.r.o., Hradec Králové
  - A-Shine, s.r.o., Pilsen
  - CLINTRIAL, s.r.o., Prague
  - FORBELI s.r.o., Prague
  - Neuropsychiatrie s.r.o., Prague
  - INEP Medical s.r.o., Prague
- Germany (9):
  - Uniklinik RWTH Aachen, Aachen
  - Charité - Universitätsmedizin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Magdeburg, Magdeburg
  - ISPG - Institut für Studien zur Psychischen Gesundheit, Mannheim
  - Technische Universität München, München
  - Universitätsklinikum Münster - Klinik für Allgemeine Neurologie, Münster
  - University Medical Center Rostock, Rostock
  - Universitätsklinikum Ulm, Ulm
- Italy (8):
  - Ospedale Bellaria - IRCCS Istituto delle Scienze Neurologiche, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - Clinica Neurologica Dipartimento di Neuroscienze e Imaging (CAST), Chieti
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS.Istituto Neurologico Carlo Besta, Milan
  - Ospedale Santa Maria della Misericordia, Perugia
  - AOU Policlinico Umberto I, Rome
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
- Netherlands (3):
  - Brain Research Center Den Bosch B.V., 's-Hertogenbosch
  - Brain Research Center Amsterdam B.V., Amsterdam
  - Brain Research Center Zwolle B.V., Zwolle
- Poland (6):
  - Revit Sp. z o.o., Podlaskie Centrum Psychogeriatrii, Bialystok
  - Krakowska Akademia Neurologii Sp. z o.o., Centrum Neurologii Klinicznej, Krakow
  - NeuroCor, ul. Medweciego 7/U12, Krakow
  - Euromedis Sp. z o.o., Centrum Medyczne EUROMEDIS, Szczecin
  - Neuroprotect Sp. z o.o., Centrum Medyczne NeuroProtect, Warsaw
  - Wielospecjalistyczne Centrum Medyczne "Ibismed" s.c., Zabrze
- Spain (5):
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Fundació ACE - Institut Català de Neurociències Aplicades, Barcelona
  - Hospital Universitario Virgen Macarena,, Seville
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Viamed Montecanal, Zaragoza

IPD SHARING:
Plan to Share IPD: No